CLINICAL TRIAL: NCT00158730
Title: Study of the Safety and Efficacy of AmBisome Loading Dose Regimen Vs. a Standard AmBisome Regimen for Initial Treatment of Invasive Aspergillosis and Other Filamentous Fungal Infections in Immunocompromised Patients
Brief Title: Study Safety/Efficacy of AmBisome Loading Dose Regimen Versus Standard AmBisome Regimen for Initial Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GS-131-101
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-11-18 (Estimated); Status verified 2005-09

CONDITIONS: Invasive Aspergillosis; Other Fungal Infections
MeSH Terms: interventions — liposomal amphotericin B

INTERVENTIONS:
Drug: AmBisome

SUMMARY:
To evaluate and compare two AmBisome dosing regimens for the initial treatment of invasive aspergillosis and other filamentous fungal infections diagnosed by modified EORTC criteria in immunocompromised patients, as determined by overall response rates at end of course of treatment.

DETAILED DESCRIPTION:
To evaluate and compare two AmBisome dosing regimens for the initial treatment of invasive aspergillosis and other filamentous fungal infections diagnosed by modified EORTC criteria in immunocompromised patients, as determined by overall response rates at end of course of treatment.

Determine and compare the following parameters for the two treatment arms:

* Safety and tolerability
* Survival rates and the rates of infection relapse at 4 weeks Post Treatment.
* Survival rate at 12 weeks after study entry.
* Time to favorable overall response and time to End of Treatment for patients with favorable overall response.
* Cumulative dose of study drug given through End of Treatment.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised due to hematologic malignancies, chemotherapy-induced neutropenia, hematopoietic stem cell transplantation, solid organ transplantation, other conditions resulting in severe neutropenia, HIV infection, prolonged corticosteroid therapy (greater than or less than 20 mg of Prednisone or equivalent for greater than or less than 3 weeks), treatment with other immunosuppressant medications, or other acquired or hereditary immunocompromising conditions that place the patients at risk for IFI. Evidence of Proven, Probably or Possible IFFI by modified EORTC criteria. Continued treatment with study drug is contingent upon confirmation of diagnosis of Proven or Probable IFI within 4 working days after study entry.

Exclusion Criteria:

* Life expectancy of less than 30 days; chronic IFI (defined as signs/symptoms of IFI present for less 4 weeks preceding entry into study;prior systemic therapy of greater than or less than 4 days with any polyene anti-fungal agent within 14 days of study enrollment;prior systemic therapy of greater than or less than 4 days with non-polyenes for the current, documented IFI. Use of another investigational, unlicensed drug within 30 days of screening or concurrent participation in another clinical trial using an investigational, unlicensed drug; serum creatinine greater than 2 x upper limit of normal (ULN), serum ALT or AST less than 5 x ULN; pregnant or lactating women; history of allergy or serious adverse reaction to any polyene anti-fungal agent.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800
Dates: Start 2003-04; Study Completion 2005-01

PRIMARY OUTCOMES:
Evaluate two regimens determined by overall response rates at end of tx.

SECONDARY OUTCOMES:
Compare Safety/tolerability; survival rates/rates of infection relapse at 4 wks post tx; survival rate at 12 wks after study entry; TOVR; time to end of tx for patients w/favorable overall response;cumulative dose

REFERENCES:
- See also: Website for AmBisome — http://www.AmBisome.com
- See also: Website for Gilead — http://www.gilead.com